CLINICAL TRIAL: NCT04929041
Title: A Randomized Phase II/III Trial of Modern Immunotherapy Based Systemic Therapy With or Without Radiation Therapy for PD-L1-Negative, Advanced Non-Small Cell Lung Cancer
Brief Title: Testing the Addition of Radiation Therapy to the Usual Treatment (Immunotherapy With or Without Chemotherapy) for Advanced Stage Non-small Cell Lung Cancer Patients Who Are PD-L1 Negative
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: End of Initial Phase of Multi-phase protocol
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-06042; NCI-2021-06042 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); A082002 (Other: Alliance for Clinical Trials in Oncology); A082002 (Other: CTEP); U10CA180821 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-06-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Adenocarcinoma; Lung Adenosquamous Carcinoma; Lung Non-Small Cell Carcinoma; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Biopsy; Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (immunotherapy, +/- chemotherapy) (Experimental): Patients receive nivolumab intravenously (IV) over 30 minutes on days 1 and 22 and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for 24 months in the absence of disease progression or unacceptable toxicity or patients may receive standard of care systemic immunotherapy. Patients also undergo MRI, CT, or PET throughout the trial. Patients may undergo blood sample collection and tissue biopsy on study as well as ECHO during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment
- Arm B (immunotherapy, +/- chemotherapy, radiation therapy) (Experimental): Patients receive 1 of 6 treatment options as in Arm A. Patients also undergo 3 fractions of radiation therapy every other day. Patients also undergo MRI, CT, or PET throughout the trial. Patients may undergo blood sample collection and tissue biopsy on study as well as ECHO during screening.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Echocardiography Test; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
  Arms: Arm B (immunotherapy, +/- chemotherapy, radiation therapy)

SUMMARY:
This phase II/III trial compares the addition of radiation therapy to the usual treatment (immunotherapy with or without chemotherapy) versus (vs.) usual treatment alone in treating patients with non-small cell lung cancer that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic) whose tumor is also negative for a molecular marker called PD-L1. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Immunotherapy with monoclonal antibodies, such as nivolumab, ipilimumab may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. The addition of radiation therapy to usual treatment may stop the cancer from growing and increase the life of patients with advanced non-small cell lung cancer who are PD-L1 negative.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess if radiation improves the progression free survival (PFS, phase II portion) and overall survival (OS, phase III portion) of advanced stage non-small cell lung cancer (NSCLC) patients with PD-L1 tumor proportion score (TPS) < 1% who receive immunotherapy with or without chemotherapy.

SECONDARY OBJECTIVES:

I. To estimate and compare the rates of >= grade 3-4 and all grade adverse events by Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0 between the arms.

II. To summarize and compare progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors (RECIST) between the arms.

III. To determine and compare the objective response rate (ORR) per RECIST between the arms (including at both irradiated and un-irradiated sites).

QUALITY OF LIFE (QOL) OBJECTIVE:

I. To assess the health-related QOL in both treatment arms.

CORRELATIVE SCIENCE OBJECTIVE:

I. To evaluate changes in the peripheral immune microenvironment between the arms.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive nivolumab intravenously (IV) over 30 minutes on days 1 and 22 and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for 24 months in the absence of disease progression or unacceptable toxicity or patients may receive standard of care systemic immunotherapy. Patients also undergo magnetic resonance imaging (MRI), computed tomography (CT), or positron emission tomography (PET) throughout the trial. Patients may undergo blood sample collection and tissue biopsy on study as well as echocardiography (ECHO) during screening.

Arm B: Patients receive nivolumab IV over 30 minutes on days 1 and 22 and ipilimumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 6 weeks for 24 months in the absence of disease progression or unacceptable toxicity or patients may receive standard of care systemic immunotherapy. Patients also undergo 3 fractions of radiation therapy every other day. Patients also undergo MRI, CT, or PET throughout the trial. Patients may undergo blood sample collection and tissue biopsy on study as well as ECHO during screening.

After completion of study treatment, patients are followed up every 3 months for 3 years and then every 6 months for years 4-5 following randomization until disease progression. Following disease progression patients are followed for survival every 6 months for up to 5 years following randomization.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of stage IV NSCLC using version American Joint Committee on Cancer (AJCC) 8th edition (includes M1a, M1b, and M1c stage disease). Patients with stage IIIB and IIIC disease are eligible if they are not a candidate for combined chemotherapy and radiation
* PD-L1 expression tumor proportion score (TPS) < 1% in tumor cells. If PD-L1 expression TPS is unevaluable or the testing could not be completed patients are not eligible. The assay must have been performed locally by a Clinical Laboratory Improvement Act (CLIA) (or equivalent) certified laboratory. The type of assay will be recorded
* For non-squamous patients only (adenocarcinoma or adenosquamous): EGFR, ALK and ROS1 testing must be done locally. No patients with known actionable EGFR mutations (except exon 20 insertion), ALK or ROS1 mutations that can be treated with oral tyrosine inhibitors
* Measurable disease based on RECIST 1.1, including at least two cancerous deposits. At least one deposit must be RECIST measurable (and not to be irradiated) while at least one OTHER deposit (measurable or non-measurable) must meet criteria for three 8 gray (Gy) doses of radiation
* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* No more than three weeks of treatment with systemic chemotherapy or immunotherapy for advanced NSCLC
* No more than three weeks of treatment with checkpoint inhibitors for metastatic lung cancer
* No treatment with chemotherapy or immunotherapy for non-metastatic disease (e.g., adjuvant therapy) within 6 months prior to registration
* No systemic immunostimulatory or immunosuppressive drugs, including > 10 mg prednisone equivalent per day, within 2 weeks or 5 half-live of the drug, whichever is shorter. Steroid premedication per local standard is allowed
* >= 1 week prior to registration since palliative (including central nervous system [CNS]) radiotherapy to any tumor site
* No prior allogeneic tissue/solid organ transplant
* No uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, uncontrolled cardiac arrhythmia, unstable angina pectoris, that would limit compliance with study requirements
* No current pneumonitis or history of non-infectious pneumonitis that required steroids
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration
* No active auto-immune disease that requires systemic therapy within 2 years prior to registration. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid release therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* No known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known hepatitis C virus (defined as HCV ribonucleic acid [RNA] [qualitative] is detected) infection
* No patients with symptomatic central nervous system metastases and/or carcinomatous meningitis. Patients with small asymptomatic brain metastases are eligible as are patients with treated brain metastases that require no steroids
* Not pregnant and not nursing, because this study involves radiation as well as potentially chemotherapy which have known genotoxic, mutagenic and teratogenic effects. Therefore, for women of childbearing potential only, a negative urine or serum pregnancy test done =< 7 days prior to registration is required
* No patients with a "currently active" second malignancy that is progressing or has required active treatment within the last 2 years. Participants with non-melanoma skin cancers or carcinoma in-situ (e.g., breast carcinoma, urothelial carcinoma or cervical cancer in situ) or localized prostate cancer (T1-3, N0, M0) that have undergone potentially curative therapy are eligible
* No hypersensitivity (>= grade 3) to immunotherapy and/or any of its excipients
* No live vaccine within 30 days prior to registration. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g.,FluMist [registered trademark]) are live attenuated vaccines and are not allowed. COVID-19 vaccine is allowed
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* Calculated (Calc.) creatinine clearance >= 45 mL/min
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) (Phase II) | From randomization to disease progression or death of all causes, whichever comes first, assessed up to 5 years
  Will be performed on an intent-to-treat (ITT) basis.
Overall survival (OS) (Phase III) | From randomization and death of all causes, assessed up to 5 years
  Will be performed on an ITT basis. The comparison of the distributions of OS between treatment arms will be done with a one-sided stratified log-rank test). The rates at various time points (e.g., every 6 months after randomization) and medians of OS for each arm will be estimated using the Kaplan-Meier estimator. The associated 95% confidence interval (CI) will be calculated using Greenwood's formula and based on a log-log transformation applied on the survival function. Hazard ratios will be estimated using a stratified Cox regression model. The final phase III analysis of OS will be considered as "positive" if the stratified log-rank test statistics Z-value greater than the critical value adjusted for type 1 error using group sequential methods. Multivariable Cox models will be used to evaluate the treatment effect on survival time and its interaction with baseline covariates, including stage, systemic therapy, histology and performance status.

SECONDARY OUTCOMES:
PFS | From randomization to disease progression or death of all causes, whichever comes first, assessed up to 5 years
  Assessed per Response Evaluation Criteria in Solid Tumors (RECIST).
Objective response rate (ORR) | Up to 5 years
  Assessed per RECIST for both irradiated and un-irradiated areas. The ORRs between treatments will be compared with Fisher's exact test. The difference of ORR between treatments will be estimated by the Miettinen-Nurminen method and its 95% CI will be given. Multivariable logistic regression will be used to evaluate the treatment effect on ORR while adjusting for significant baseline covariates.
Quality of life | Up to 5 years
Incidence of treatment-related adverse events | Up to 5 years
  Treatment-related toxicity will be summarized by grade, type, and system organ class. Comparisons of the percentages of patients experiencing an adverse event between Arm A and Arm B will be performed using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Bestvina, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (170):
- United States (170):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Providence Queen of The Valley, Napa, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - City of Hope Upland, Upland, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - CTCA at Southeastern Regional Medical Center, Newnan, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Waukee Clinic, Waukee, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - The Iowa Clinic PC, West Des Moines, Iowa
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Manhattan Eye Ear and Throat Hospital, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Upstate Cancer Center at Hill Radiation Oncology, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Health Tappahannock Hospital, Tappahannock, Virginia
  - Legacy Cancer Institute Medical Oncology and Day Treatment, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Schild SE, Wang X, Bestvina CM, Williams T, Masters G, Singh AK, Stinchcombe TE, Salama JK, Wolf S, Zemla T, Duma N, Chun SG, Amini A, Kozono D, Watt C. Alliance A082002 -a randomized phase II/III trial of modern immunotherapy-based systemic therapy with or without SBRT for PD-L1-negative, advanced non-small cell lung cancer. Clin Lung Cancer. 2022 Jul;23(5):e317-e320. doi: 10.1016/j.cllc.2022.04.004. Epub 2022 Apr 30. PMID 35613998